CLINICAL TRIAL: NCT01505764
Title: The Role of Ghrelin in Cancer Cachexia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Helsinn Therapeutics (U.S.), Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-013-08F; HT-ANAM-208 (Other: Helsinn Therapeutics (U.S.), Inc)
Record Dates: First submitted 2011-12-07; First posted 2012-01-09 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Cancer Cachexia
Keywords: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Anamorelin HCl) (Experimental): Anamorelin HCl
  Interventions: Drug: Anamorelin HCl
- Arm 2 (Placebo) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anamorelin HCl — 100 mg tablets; oral administration every day for 84 days, at least 1 hour before the first meal of the day.
  Arms: Arm 1 (Anamorelin HCl)
Drug: Placebo — Placebo tablets identical in appearance to active tablets; oral administration once a day for 84 days, at least 1 hour before the first meal of the day.
  Arms: Arm 2 (Placebo)

SUMMARY:
Cancer is often coupled with a condition called cachexia. In this condition, individuals continue to lose weight and lean body mass, which means their muscles are getting smaller and weaker. Studies have shown that cancer patients who are losing weight often are responding poorly to chemotherapy, are at greater risk of infection and have a reduced life expectancy. Also, people may not want to eat. To date, there are no approved treatments available for this condition.

This study is going to study the benefits of the use of the study drug, Anamorelin hydrochloride (HCl) in treatment or prevention of cachexia associated with cancer. Studies done before with the study drug have shown that the drug can help the cachectic condition. The purpose of this research study is to evaluate the effectiveness of Anamorelin HCl compared to placebo on body composition (amount of cell mass, fat, muscle, etc.) including measurements of body potassium and nitrogen stores.

In addition to the above, the study will also assess the effect of the study drug on handgrip strength, body weight, lean muscle mass, quality of life, appetite & food intake, certain blood markers, energy expenditure (the amount of energy participants burn), functional performance, safety and tolerability of Anamorelin HCl.

DETAILED DESCRIPTION:
Subjects enrolled in the study will be randomly chosen to receive either Anamorelin HCL at a dose of 100 mg per day for 12 weeks or matching placebo. The chances of receiving anamorelin or placebo are 1 in 2. Which subject receives anamorelin or placebo will be decided at random. Neither the subject nor the study doctor will know which study drug the subject is receiving. The subject will be asked to visit the clinic at Day 1, Day 28, Day 56 and Day 84. There will also be a Day 112 follow-up visit and the medical records will be checked after that to see how the subjects are doing.

ELIGIBILITY:
Inclusion Criteria:

* Must have incurable, histologically or cytologically documented Non-Small Cell Lung Cancer or Colo-rectal Cancer.
* Females and males at least 18 years of age.
* Documented histologic or cytologic diagnosis of American Joint Committee on Cancer (AJCC) unresectable Stage III or IV NSCLC and/or stage III or IV colorectal cancer (CRC) (not amenable to curative resection).
* Involuntary weight loss of 5% body weight over a period of 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 2 at screening.
* Estimated life expectancy of greater than 4 months at the time of screening.
* Presence and functional use of both hands.
* Able to understand and comply with the procedures of the handgrip strength evaluation.
* If the patient is a woman of childbearing potential or a fertile man, he/she must agree to use an effective form of contraception during the study and for 28 days following the last dose of study medication.
* Willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures.

Exclusion Criteria:

* Other forms of lung cancer.
* Women who are pregnant or breast-feeding.
* Obesity.
* Recent active excessive alcohol or illicit drug use current use of marijuana or history of marijuana use over the previous 6 months.
* Severe depression.
* Other causes of cachexia such as:

  * Liver disease (AST or ALT > 3x normal levels)
  * Renal failure (creatinine > 2.5 mg/dL)
  * Untreated thyroid disease
  * Class III-IV CHF
  * AIDS
  * Other cancer diagnosed within the past five years other than non-melanoma skin cancer and prostate cancer
  * Severe COPD requiring use of home O2.
* Inability to increase food intake.
* Recent administration of highly emetogenic chemotherapy.
* Known HIV, active hepatitis B or C (with increased LFTs), or active tuberculosis.
* Patients who have received two prior regimens of cytotoxic chemotherapy and are undergoing, or planning to undergo, a third regimen of cytotoxic chemotherapy.
* Currently taking prescription medications intended to increase appetite or treat weight loss; these include, but are not limited to:

  * Testosterone
  * Androgenic compounds
  * Megestrol acetate
  * Methylphenidate
  * Dronabinol
* Current use of steroids or history of use over the previous 6 months except as pre- and post-medications for chemotherapy administration.
* Patients unable to readily swallow oral tablets.
* An active, uncontrolled infection.
* Uncontrolled diabetes mellitus.
* Known or suspected brain metastases.
* Patients receiving strong CYP3A4 inhibitors.
* Patients receiving tube feedings or parenteral nutrition.
* Patients with any concomitant medical or psychiatric condition or social situation that would make it difficult to comply with protocol requirements, including the inability to comply with handgrip strength determinations in both hands; for example, pre-existing neurological impairment.
* Previous exposure to Anamorelin HCl.
* Patients actively receiving a concurrent investigational agent, or any patients that have received an investigational agent within four weeks prior to randomization.
* Current use of diuretics or history of intermittent diuretic usage for any reason over the previous 3 months.
* History of claustrophobia.
* Cachexia deemed by the investigator to be solely due to chemo or radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M. Garcia, MD PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects were consented, 9 received drug or placebo, 5 completed the study.
Period: Overall Study
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Started | 6 | 3
Completed (not completed due to poor recruitment) | 3 | 2
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo) | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: years] | 56 [48 to 72] | 58 [56 to 73] | 57 [48 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Body Potassium.
Description: percentage change from baseline
Time Frame: day 84
Population: cancer cachexia patients
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 3 | 2
percentage change | -2.13 (5.48) | -0.72 (2.11)

2. Secondary Outcome: Lean Mass Measured by Densitometry.
Description: lean body mass measured by DEXA. Percentage of change day 84-baseline.
Time Frame: day 84
Population: only two subjects in each group completed this measure.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 2 | 2
percentage change | 2.12 (3.05) | -1.44 (0.5)

3. Secondary Outcome: Muscle Strength as Measured by Grip Strength.
Description: Dominant hand grip strength day 84 - percent change from baseline
Time Frame: day 84
Population: Cancer cachexia patients
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 3 | 2
percentage change | 0.31 (11.19) | -10.45 (14.49)

4. Secondary Outcome: Body Weight.
Description: percent change from day 84-baseline
Time Frame: day 84
Population: cancer cachexia patients
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 3 | 2
percentage change | 1.7 (3.19) | -1.8 (0.07)

5. Secondary Outcome: Quality of Life.
Description: Quality of life as assessed using the FACIT-F Patient Reported Outcome assessments - percentage of change day 84-baseline
Time Frame: day 84
Population: cancer cachexia patients
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 3 | 2
percentage change | -6.54 (4.9) | -14.32 (3.78)

6. Secondary Outcome: Appetite.
Description: Appetite measured by a visual analogue scale ASAS. Percentage of change day84-baseline
Time Frame: day 84
Population: cancer cachexia patients
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 3 | 2
percentage change | 8.33 (38.18) | 1.66 (25.92)

7. Secondary Outcome: Resting Energy Expenditure.
Description: % change between day 84 and baseline
Time Frame: day 84
Population: cancer cachexia patients
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 3 | 2
percentage change | -1.02 (13.8) | -2.58 (2.75)

8. Secondary Outcome: Functional Performance.
Description: Functional performance using stair-climbing power day 84 percent change from baseline
Time Frame: day 84
Population: only two subjects in each group completed this measure.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 2 | 2
percentage change | 22.53 (9.87) | -13.8 (12.36)

9. Secondary Outcome: Body Composition.
Description: Body composition as measured by Total body nitrogen. Percentage of change day 84-baseline
Time Frame: day 84
Population: only two subjects in each group completed this outcome
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 2 | 2
percentage change | -5.7 (3.4) | 6.31 (4.2)

10. Secondary Outcome: Stair Climbing Power
Description: Percent change from baseline
Time Frame: day 84
Population: only two subjects in each group completed this outcome
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 2 | 2
percentage change | -30.39 (27.86) | 4.12 (15.23)

11. Secondary Outcome: 1-repetition Max. Strength
Description: leg extension - percentage of change day 84 to baseline
Time Frame: day 84
Population: only two subjects in each group completed this outcome
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 2 | 2
percentage change | 93.87 (70.53) | -8.29 (0.56)

12. Secondary Outcome: Food Diary Calorie Count
Description: change between day 84 and baseline
Time Frame: day 84
Population: cancer cachexia patients
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Number analyzed (Participants) | 3 | 2
percentage change | -21 (14) | -12 (19)

ADVERSE EVENTS:
Arm/Group | Arm 1 (Anamorelin HCl) | Arm 2 (Placebo)
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/4
Other Adverse Events (participants affected / at risk) | 2/6 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Anamorelin HCl) (N=6) | Arm 2 (Placebo) (N=4)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Anamorelin HCl) (N=6) | Arm 2 (Placebo) (N=4)
pain (Nervous system disorders) | 1 (1) | 0 (0)
fatigue (Nervous system disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No